CLINICAL TRIAL: NCT06400277
Title: In-Vivo Comparison of Different Impression Methods in Complete Edentulous Upper Jaw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sinem Kahya Karaca, Research Assistant, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KA-22026
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Edentulous Jaw
Keywords: Edentulous Jaw; Digital Impression; Physical Impression
MeSH Terms: conditions — Jaw, Edentulous | interventions — Denture, Complete

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Irreversible Hydrocolloid (Other): Final impression taken with irreversible hydrocolloid impression material and stock tray in single step.
  Interventions: Other: Edentulous maxilla final impression for complete denture
- Zinc Oxide Eugenol (Other): Final impression taken with zinc oxide eugenol impression material and individual tray in two steps.
  Interventions: Other: Edentulous maxilla final impression for complete denture
- Intraoral Scanner - Artificial Intelligence Off (Other): Final impression taken with intraoral scanner in artificial intelligence mode deactivated in single step.
  Interventions: Other: Edentulous maxilla final impression for complete denture
- Intraoral Scanner - Artificial Intelligence On (Other): Final impression taken with intraoral scanner in artificial intelligence mode activated in single step.
  Interventions: Other: Edentulous maxilla final impression for complete denture
- Intraoral Scanner - Modified (Other): Final impression taken with intraoral scanner in two steps using occlusal rim.
  Interventions: Other: Edentulous maxilla final impression for complete denture

INTERVENTIONS:
Other: Edentulous maxilla final impression for complete denture — Final impressions of edentulous maxilla separated in two groups. In physical impression group stock and individual trays and physical impression materials used.

SUMMARY:
In this study, it was aimed to compare the impressions taken with different impression techniques for the production of tissue-supported complete dentures from individuals with complete edentulous upper jaws. For this purpose, 15 individuals with complete edentulism in the upper jaw were asked to participate in the study. In addition to agreeing to participate in the study after reading the consent form, these individuals should have been using tissue-supported complete dentures in the upper jaw for at least 3 months. They should also have healthy mucosa without local factors such as tissue hyperplasia, atrophic crests, allergic reaction, epulis fissuratum. A total of five final impressions will then be taken from these individuals in two sessions. Two of these impressions will be obtained with the traditional method and three with the digital method. The traditional impression group will include one-step (ALG) and two-step (ZOE) impression techniques. The digital impression group will include the digital impression taken when the artificial intelligence is deactivated (A.I OFF), the digital impression taken when the artificial intelligence is activated (A.I ON) and the modified technique (MOD). In the first appointment, the first impressions will be taken for the traditional and digital groups. Intraoral exclusion and isolation will be provided before the digital first impression. With the A.I mode of the intraoral scanner (TRIOS4; 3Shape A/S, Copenhagen, Denmark) deactivated, scanning will be performed in accordance with the scanning protocol recommended by the company. A metal stock tray suitable for the dental arch will then be selected for the preliminary impression of the traditional impression group. The impression will be taken in one step with irreversible hydrocolloid impression material. The impression will be digitized with the same intraoral scanner within the first 10 minutes after impression taking. Both impressions will be digitally transferred to the dental laboratory as stl data. Using computer aided design (CAD) software (Exocad DentalCAD 2.4 Plovdiv), an individual tray will be designed for the ZOE impression in the traditional group and a pedestal for the MOD impression in the digital impression group. The designs will be transferred to the computer aided manufacturing (CAM) unit and produced with a 3D printer using dental resin. The occlusal-rim (OR) will be prepared by adding wax on the base.

In the second appointment, the cheek and lips will be excluded in the same way before scanning. For A.I OFF and A.I ON, recordings will be taken when the artificial intelligence is deactivated and activated, respectively. Then, occlusal vertical dimension, intermaxillary relationship and aesthetic parameters will be determined with OR before scanning for the MOD group. Reference areas will be created on the buccal and palatinal walls to facilitate scanning of the OR. To avoid retention problems during scanning, a silicone-based impression material with a fluid consistency will be applied to the tissue surface of the OR and placed in the mouth. Scanning will be performed according to the protocol proposed by Lo Russo et al. For the traditional impression group, the ALG impression will be taken with a metal stock tray using irreversible hydrocolloid impression material in a single step. The impression will be digitized with an intraoral scanner within ten minutes of completion. Then, the edges of the individual tray for ZOE will be shaped with impression compound to ensure peripheral closure. The impression will be completed with zinc-oxide eugenol impression material. The impression will be digitized. These measurements will then be compared using a reverse-engineering program (Geomagic design X version 2016.1.0, 3D Systems Inc. Rock Hill, SC). Before the comparison, in the same program, the parts to be evaluated on the ZOE in the conventional group and A.I OFF in the digital group will be divided into regions. These areas will be divided into four sections as right and left vestibular region, postdam area, hard palate region, except for the A.I OFF-MOD comparison group. In the A.I OFF-MOD comparison group, it will include the right and left initial areas, including the areas where scanning starts in the second scan of the MOD method. In addition, all measurements will be compared in terms of the whole surface and all measurement boundaries including the whole measurement surface as one. The comparison groups are ZOE-ALG, ZOE-A.I OFF, A.I OFF-A.I ON, A.I OFF-MOD. The measurements in the comparison groups will be overlapped first with the initial alignment and then with the best fit alignment algorithm. All sections will be evaluated individually with the "3D compare" feature and the amount of deviation in the areas to be evaluated will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who had been using maxillary complete denture for at least 3 months
* Volunteers were clinically evaluated for healthy oral mucosa

Exclusion Criteria:

* Volunteers who had general health problems
* Volunteers who had of tissue hyperplasia, labile alveolar crest, allergic reaction to the prosthesis, percussion or mucosal irritation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Three Dimensional Difference Between Irreversible Hydrocolloid and Zinc Oxide Eugenol Impressions | Through study completion, an average of 6 months
  Evaluation of the three-dimensional difference between two impressions using a reverse-engineering program and quantification of the deviation
Three Dimensional Difference Between Zinc Oxide Eugenol and Intraoral Scanner AI Off Impressions | Through study completion, an average of 6 months
  Evaluation of the three-dimensional difference between two impressions using a reverse-engineering program and quantification of the deviation
Three Dimensional Difference Between Intraoral Scanner AI Off and AI On Impressions | Through study completion, an average of 6 months
  Evaluation of the three-dimensional difference between two impressions using a reverse-engineering program and quantification of the deviation
Three Dimensional Difference Between Intraoral Scanner AI Off and Modified Impressions | Through study completion, an average of 6 months
  Evaluation of the three-dimensional difference between two impressions using a reverse-engineering program and quantification of the deviation

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Kahya Karaca, Principal Investigator — Hacettepe University; Kıvanç Akça, Prof. Dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lo Russo L, Salamini A, Troiano G, Guida L. Digital dentures: A protocol based on intraoral scans. J Prosthet Dent. 2021 Apr;125(4):597-602. doi: 10.1016/j.prosdent.2020.02.006. Epub 2020 Apr 21. PMID 32331785
- [Background] Lo Russo L, Caradonna G, Troiano G, Salamini A, Guida L, Ciavarella D. Three-dimensional differences between intraoral scans and conventional impressions of edentulous jaws: A clinical study. J Prosthet Dent. 2020 Feb;123(2):264-268. doi: 10.1016/j.prosdent.2019.04.004. Epub 2019 May 29. PMID 31153614
- [Background] Chebib N, Kalberer N, Srinivasan M, Maniewicz S, Perneger T, Muller F. Edentulous jaw impression techniques: An in vivo comparison of trueness. J Prosthet Dent. 2019 Apr;121(4):623-630. doi: 10.1016/j.prosdent.2018.08.016. Epub 2018 Dec 21. PMID 30580982
- [Derived] Kahya Karaca S, Akca K. Comparison of conventional and digital impression approaches for edentulous maxilla: clinical study. BMC Oral Health. 2024 Nov 14;24(1):1378. doi: 10.1186/s12903-024-05151-3. PMID 39543593

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT06400277/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT06400277/ICF_001.pdf